CLINICAL TRIAL: NCT03568721
Title: Postoperative Effects of Chewing Gum, Ibuprofen and Acetaminophen on Pain After Initial Archwire Placement: a Randomized Controlled Trial
Brief Title: Postoperative Effects of Chewing Gum, Ibuprofen and Acetaminophen on Pain After Initial Archwire Placement
Acronym: PECI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Diego Junior da Silva Santos, DDS,MsD, Principal Investigator, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 173112
Record Dates: First submitted 2018-06-02; First posted 2018-06-26 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Pain
Keywords: pain; orthodontics
MeSH Terms: conditions — Pain | interventions — Ibuprofen; GDF15 protein, human; Acetaminophen; Chewing Gum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ibuprofen (Experimental): ibuprofen (400 mg) immediately after insertion of the initial archwire and 6/6 hs for a week if there is any orthodontic pain.
  Interventions: Drug: Ibuprofen
- acetaminophen (Experimental): acetaminophen (500 mg) immediately after insertion of the initial archwire and 6/6 hs for a week if there is any orthodontic pain.
  Interventions: Drug: Acetaminophen
- chewing gum (Experimental): chewing gum (01 tablet) immediately after insertion of the initial archwire and 6/6 hs of chewing gum for a week if there is any orthodontic pain.
  Interventions: Other: Chewing gum
- control (No Intervention): control (no reliever for orthodontic pain)

INTERVENTIONS:
Drug: Ibuprofen — prescription of ibuprofen 400 mg
  Other Names: non steroidal drug
  Arms: ibuprofen
Drug: Acetaminophen — prescription of acetaminophen 500 mg
  Other Names: paracetamol
  Arms: acetaminophen
Other: Chewing gum — prescription of one tablet of chewing gum
  Arms: chewing gum

SUMMARY:
The purpose of this study is to compare the efficacy of ibuprofen, acetaminophen, chewing gum in reducing orthodontic pain. This study include 81 patients to be classified into 4 groups of 19 each: ibuprofen (400 mg), acetaminophen (500 mg), chewing gum and control. The patients in each group will receive 1 method immediately after placement of the initial archwire and every 6 hours for a week if they experiences pain. Pain perception will be recorded by the patients while jaw rest position and fitting back teeth at 2 hours, 24 hours, 2 days, 3 days, 7 days and 21 days after archwire placement, using a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* moderate teeth crowding
* no need for tooth extraction to orthodontic reasons

Exclusion Criteria:

* presence of autoimmune diseases
* history of orthodontic treatment with fixed appliances

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2015-01-25 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Orthodontic pain measurement by marking 100 millimeters visual analogue scales. | 2 hours, 24 hours, 2 days, 3 days, 7 days and 21 days after archwire placement.
  to compare the efficacy of ibuprofen, acetaminophen and chewing gum in changing orthodontic pain by marking in between two points in a 100 millimeters visual analogue scale that starts from the left (no pain) and end to the right (exacerbated pain) at different time points.

SECONDARY OUTCOMES:
Chewing gum as a non pharmacologic alternative for orthodontic pain control by marking 100 millimeters visual analogue scales. | 2 hours, 24 hours, 2 days, 3 days, 7 days and 21 days after archwire placement.
  to verify if chewing gum can be a non-pharmacologic method for orthodontic pain control by marking in between two points in a 100 millimeters visual analogue scale that starts from the left (no pain) and ends to the right (exacerbated pain) at different time points.
Pain at rest X fitting back teeth by marking 100 millimeters visual analogue scales. | 2 hours, 24 hours, 2 days, 3 days, 7 days and 21 days after archwire placement.
  to verify wich group has less pain and if in rest or in fitting back teeth by marking in between two points in a 100 millimeters visual analogue scale that starts from the left (no pain) and end to the right (exacerbated pain) at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: DIEGO J SANTOS, MSc, Principal Investigator — Rio de Janeiro State University; JONAS CAPELLI, PhD, Study Director — Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farzanegan F, Zebarjad SM, Alizadeh S, Ahrari F. Pain reduction after initial archwire placement in orthodontic patients: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2012 Feb;141(2):169-73. doi: 10.1016/j.ajodo.2011.06.042. PMID 22284284
- [Background] Sandhu SS, Sandhu J. Orthodontic pain: an interaction between age and sex in early and middle adolescence. Angle Orthod. 2013 Nov;83(6):966-72. doi: 10.2319/030113-174.1. Epub 2013 May 24. PMID 23705940
- [Background] Angelopoulou MV, Vlachou V, Halazonetis DJ. Pharmacological management of pain during orthodontic treatment: a meta-analysis. Orthod Craniofac Res. 2012 May;15(2):71-83. doi: 10.1111/j.1601-6343.2012.01542.x. PMID 22515183
- [Background] Bergius M, Berggren U, Kiliaridis S. Experience of pain during an orthodontic procedure. Eur J Oral Sci. 2002 Apr;110(2):92-8. doi: 10.1034/j.1600-0722.2002.11193.x. PMID 12013568
- [Background] Erdinc AM, Dincer B. Perception of pain during orthodontic treatment with fixed appliances. Eur J Orthod. 2004 Feb;26(1):79-85. doi: 10.1093/ejo/26.1.79. PMID 14994886
- [Background] Canavarro C, Teles RP, Capelli Junior J. Matrix metalloproteinases -1, -2, -3, -7, -8, -12, and -13 in gingival crevicular fluid during orthodontic tooth movement: a longitudinal randomized split-mouth study. Eur J Orthod. 2013 Oct;35(5):652-8. doi: 10.1093/ejo/cjs053. Epub 2012 Sep 17. PMID 22989715
- [Background] Davies GM, Worthington HV, Ellwood RP, Blinkhorn AS, Taylor GO, Davies RM, Considine J. An assessment of the cost effectiveness of a postal toothpaste programme to prevent caries among five-year-old children in the North West of England. Community Dent Health. 2003 Dec;20(4):207-10. PMID 14696738
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720
- [Background] Hwang JY, Tee CH, Huang AT, Taft L. Effectiveness of thera-bite wafers in reducing pain. J Clin Orthod. 1994 May;28(5):291-2. No abstract available. PMID 8613507
- [Background] White LW. Pain and cooperation in orthodontic treatment. J Clin Orthod. 1984 Aug;18(8):572-5. No abstract available. PMID 6595271
- [Background] Krishnan V, Davidovitch Z. The effect of drugs on orthodontic tooth movement. Orthod Craniofac Res. 2006 Nov;9(4):163-71. doi: 10.1111/j.1601-6343.2006.00372.x. PMID 17101023
- [Background] Simmons KE, Brandt M. Control of orthodontic pain. J Indiana Dent Assoc. 1992 Jul-Aug;71(4):8-10. PMID 1432346
- [Background] Keith DJ, Rinchuse DJ, Kennedy M, Zullo T. Effect of text message follow-up on patient's self-reported level of pain and anxiety. Angle Orthod. 2013 Jul;83(4):605-10. doi: 10.2319/091812-742.1. Epub 2012 Dec 4. PMID 23210546
- [Background] Brown DF, Moerenhout RG. The pain experience and psychological adjustment to orthodontic treatment of preadolescents, adolescents, and adults. Am J Orthod Dentofacial Orthop. 1991 Oct;100(4):349-56. doi: 10.1016/0889-5406(91)70073-6. PMID 1927986
- [Background] Bergius M, Broberg AG, Hakeberg M, Berggren U. Prediction of prolonged pain experiences during orthodontic treatment. Am J Orthod Dentofacial Orthop. 2008 Mar;133(3):339.e1-8. doi: 10.1016/j.ajodo.2007.09.013. PMID 18331926
- [Background] Scheurer PA, Firestone AR, Burgin WB. Perception of pain as a result of orthodontic treatment with fixed appliances. Eur J Orthod. 1996 Aug;18(4):349-57. doi: 10.1093/ejo/18.4.349. PMID 8921656
- [Background] Bernhardt MK, Southard KA, Batterson KD, Logan HL, Baker KA, Jakobsen JR. The effect of preemptive and/or postoperative ibuprofen therapy for orthodontic pain. Am J Orthod Dentofacial Orthop. 2001 Jul;120(1):20-7. doi: 10.1067/mod.2001.115616. PMID 11455373
- [Background] Jones M, Chan C. The pain and discomfort experienced during orthodontic treatment: a randomized controlled clinical trial of two initial aligning arch wires. Am J Orthod Dentofacial Orthop. 1992 Oct;102(4):373-81. doi: 10.1016/0889-5406(92)70054-e. PMID 1456222
- [Background] Cioffi I, Piccolo A, Tagliaferri R, Paduano S, Galeotti A, Martina R. Pain perception following first orthodontic archwire placement--thermoelastic vs superelastic alloys: a randomized controlled trial. Quintessence Int. 2012 Jan;43(1):61-9. PMID 22259810
- [Background] Salmassian R, Oesterle LJ, Shellhart WC, Newman SM. Comparison of the efficacy of ibuprofen and acetaminophen in controlling pain after orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):516-21. doi: 10.1016/j.ajodo.2007.05.020. PMID 19361739
- [Background] Patel S, McGorray SP, Yezierski R, Fillingim R, Logan H, Wheeler TT. Effects of analgesics on orthodontic pain. Am J Orthod Dentofacial Orthop. 2011 Jan;139(1):e53-8. doi: 10.1016/j.ajodo.2010.07.017. PMID 21195257